CLINICAL TRIAL: NCT01586988
Title: A Parenting Intervention for HIV+ Moms: The IMAGE Program
Brief Title: A Parenting and Self-Care Intervention for HIV Infected Mothers
Acronym: IMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R01MH086329 (NIH); R01MH086329 (NIH)
Record Dates: First submitted 2011-07-01; First posted 2012-04-27 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: HIV
Keywords: HIV; Parenting; self-care; disclosure; medication adherence; mother; child; adolescent
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMAGE Intervention (Experimental): mothers are provided the IMAGE Parenting and Self-Care intervention
  Interventions: Behavioral: IMAGE Intervention
- Control (No Intervention): Standard care.

INTERVENTIONS:
Behavioral: IMAGE Intervention — Mothers in the intervention will receive four individual intervention sessions with a facilitator. The sessions will cover parenting and self care skills.
  Arms: IMAGE Intervention

SUMMARY:
The IMAGE intervention was developed to improve parenting and self-care skills in mothers infected with HIV. It is expected that an improvement in these areas will in turn improve the mother's physical and mental health as well as the child's mental health and behavioral adjustment.

DETAILED DESCRIPTION:
Worldwide, close to half the adults living with HIV are women and a large proportion of these women are of child-bearing age. Whereas anyone living with HIV faces the physical challenges of living with a chronic disease, as well as the material and social impact of the stigma associated with the disease, mothers living with HIV must also meet the demands of childrearing while mitigating the negative impact of the disease upon their family. Mothers with HIV report that this is their greatest source of stress. Moreover, children of these mothers, growing up with a parent with a chronic, stigmatized, and often fatal disease, are considered a high-risk group. The IMAGE intervention was designed to improve parenting and self-care skills in mothers with HIV in order to improve the mother's physical and mental health as well as the child's mental health and behavioral adjustment.

ELIGIBILITY:
Inclusion Criteria:

* mother has confirmed diagnosis of HIV
* well (HIV-) child, 6 to 14 years of age
* mother is English or Spanish speaking
* child is English speaking

Exclusion Criteria:

* low cognitive/intellectual functioning (<75) in mother or child
* psychosis in mother or child

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Targeted Behaviors, Practices, and Skills and Maternal and Child Health | 3-months, 6-months, and 12-months
  Specific targets of the intervention, including parenting practices, parenting behaviors, and self care skills, will be evaluated. In addition, the mother's physical and mental health and the child's mental health and behavioral adjustment will be evaluated.

SECONDARY OUTCOMES:
Parenting Self-efficacy | 3-months, 6-months, and 12-months
  Perceptions of effectiveness in the parental role and general parenting self-efficacy will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Isap, Los Angeles, California, United States

REFERENCES:
- [Result] Murphy DA, Armistead L, Payne DL, Marelich WD, Herbeck DM. Pilot trial of a parenting and self-care intervention for HIV-positive mothers: the IMAGE program. AIDS Care. 2017 Jan;29(1):40-48. doi: 10.1080/09540121.2016.1204416. Epub 2016 Jul 4. PMID 27377577